CLINICAL TRIAL: NCT02222207
Title: A Combined Phase IIa / IIb Study of the Efficacy, Safety, and Tolerability of Repeated Topical Doses of Regorafenib Eye Drops, in Treatment-naïve Subjects With Neovascular Age Related Macular Degeneration
Brief Title: Regorafenib Eye Drops: Investigation of Efficacy and Safety in Neovascular Age Related Macular Degeneration
Acronym: DREAM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15984; 2012-003763-22 (EudraCT Number)
Record Dates: First submitted 2014-08-20; First posted 2014-08-21 (Estimated); Results first posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-07

CONDITIONS: Macular Degeneration
Keywords: neovascular Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — regorafenib; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Regorafenib [A] (Experimental): Part A: Patients will receive Regorafenib eye drops
  Interventions: Drug: Regorafenib, ophthalmic oily suspension (BAY73-4506)
- Regorafenib [B1] (Experimental): Part B: Regorafenib eye drops dose 1; plus sham IVT (Intravitreal therapy) once every 4 weeks
  Interventions: Drug: Regorafenib, ophthalmic oily suspension (BAY73-4506); Procedure: Sham IVT
- Regorafenib [B2] (Experimental): Part B: Regorafenib eye drops dose 2; plus sham IVT (Intravitreal therapy) once every 4 weeks
  Interventions: Drug: Regorafenib, ophthalmic oily suspension (BAY73-4506); Procedure: Sham IVT
- Regorafenib [B3] (Experimental): Part B: Regorafenib eye drops dose 3; plus sham IVT (Intravitreal therapy) once every 4 weeks
  Interventions: Drug: Regorafenib, ophthalmic oily suspension (BAY73-4506); Procedure: Sham IVT
- Regorafenib [B4] (Experimental): Part B: Regorafenib eye drops dose 4; plus sham IVT (Intravitreal therapy) once every 4 weeks
  Interventions: Drug: Regorafenib, ophthalmic oily suspension (BAY73-4506); Procedure: Sham IVT
- Regorafenib [B5] (Experimental): Part B: Regorafenib eye drops dose 5; plus sham IVT (Intravitreal therapy) once every 4 weeks
  Interventions: Drug: Regorafenib, ophthalmic oily suspension (BAY73-4506); Procedure: Sham IVT
- Regorafenib [B6] (Experimental): Part B: Regorafenib eye drops dose 6; plus sham IVT (Intravitreal therapy) once every 4 weeks
  Interventions: Drug: Regorafenib, ophthalmic oily suspension (BAY73-4506); Procedure: Sham IVT
- Ranibizumab (Active Comparator): Ranibizumab IVT once every 4 weeks; plus placebo eye drops to match the regorafenib eye drop regimens
  Interventions: Drug: Ranibizumab; Drug: Placebo

INTERVENTIONS:
Drug: Regorafenib, ophthalmic oily suspension (BAY73-4506) — Subjects receive Regorafenib as eye drops
  Arms: Regorafenib [A]; Regorafenib [B1]; Regorafenib [B2]; Regorafenib [B3]; Regorafenib [B4]; Regorafenib [B5]; Regorafenib [B6]
Procedure: Sham IVT — Sham injections
  Arms: Regorafenib [B1]; Regorafenib [B2]; Regorafenib [B3]; Regorafenib [B4]; Regorafenib [B5]; Regorafenib [B6]
Drug: Ranibizumab — Subjects receive Ranibizumab as intravitreal injection
  Arms: Ranibizumab
Drug: Placebo — Placebo eye drops
  Arms: Ranibizumab

SUMMARY:
Part A (Phase IIa):

Primary objectives:

The study part A is designed to investigate whether the use of regorafenib eye drops can help patients with neovascular (wet) Age-Related Macular Degeneration (wAMD) to see better after 4 weeks and 12 weeks after inclusion into this study.

Secondary objectives:

The study will also evaluate the safety and tolerability of the regorafenib eye drops.

Part B (Phase IIb):

Primary objectives:

The study part B is designed to investigate:

* how often the regorafenib eye drops need to be given per day
* whether the use of regorafenib eye drops can help patients with neovascular (wet) Age-Related Macular Degeneration (wAMD) to see better after 4 weeks and 12 weeks after inclusion into this study.

Secondary objectives:

The study will also evaluate how the different dosings of regorafenib eye drops affect patients vision, the safety and the tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Able to read (or, if unable to read due to visual impairment, be read to verbatim by the person administering the informed consent or a family member) and able to understand the informed consent form (ICF)
* Men and women ≥ 50 years of age
* Active primary subfoveal CNV (Choroidal neovascularization) lesions secondary to AMD (Age-related macular degeneration), including juxtafoveal lesions that affect the fovea as evidenced by FA (Fluorescein angiography) in the study eye and reviewed by the central reading center
* The area of CNV must occupy at least 50% of total lesion in the study eye, as determined by FA review at the central reading center
* Evidence of intraretinal and/or subretinal fluid on OCT (Optical coherence tomography)
* Early Treatment Diabetic Retinopathy Study BCVA of 73 to 25 letters (20/40 to 20/320 Snellen equivalent) in the study eye
* Willing, committed, and able to return for all clinic visits and complete all study related procedures
* Women of childbearing potential and men must agree to use adequate contraception when sexually active. This applies since signing of the ICF until one month after the EOS (end of study) visit. The definition of adequate contraception will be based on the judgment of the investigator.

Exclusion Criteria:

* Concurrent disease in the study eye, other than AMD (e.g., corneal diseases and dystrophies, conjunctival diseases, eye lid abnormalities, or any other diseases of the cornea and macula, or optic nerve abnormality) that could compromise visual acuity, likely require medical or surgical intervention during the study period, would limit the potential to gain or lose vision during study treatment, or could otherwise confound interpretation of the results
* Total lesion size (including neovascularization, scar, blood) > 12 disc areas (30.5 mm2) as assessed by FA
* Only one functional eye, even if that eye is otherwise eligible for the study
* Prior ocular or systemic treatment or surgery for neovascular AMD in the study eye except dietary supplements or vitamins
* Prior treatment with any systemic anti-VEGF (Vascular endothelial growth factor) agent
* Use of systemic or ocular treatment with an investigational drug within 12 weeks prior to start of study treatment
* Any other condition that would require frequent chronic co-administration of other topical eye medications that would interfere with study drug administration (e.g. contact lens)
* Symptoms or conditions consistent with contraindications listed in the current local label for ranibizumab
* Participation in an investigational study within 30 days prior to start of study treatment that involved treatment with any drug (excluding vitamins and minerals) or device
* Lactating women and women of child-bearing potential with either a positive pregnancy test result or no pregnancy test at screening are excluded. Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (132):
- United States (37):
  - Tucson, Arizona
  - Arcadia, California
  - Beverly Hills, California
  - Campbell, California
  - Costa Mesa, California
  - Laguna Hills, California
  - Mountain View, California
  - Santa Ana, California
  - Golden, Colorado
  - Boynton Beach, Florida
  - Fort Myers, Florida
  - Miami, Florida
  - Plantation, Florida
  - Sarasota, Florida
  - Stuart, Florida
  - Winter Haven, Florida
  - Decatur, Georgia
  - New Albany, Indiana
  - Leawood, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Eunice, Louisiana
  - Boston, Massachusetts
  - Grand Rapids, Michigan
  - Florissant, Missouri
  - Teaneck, New Jersey
  - Asheville, North Carolina
  - West Mifflin, Pennsylvania
  - Greenville, South Carolina
  - Rapid City, South Dakota
  - Austin, Texas
  - Houston, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - Temple, Texas
  - The Woodlands, Texas
  - Charlottesville, Virginia
- Australia (5):
  - Strathfield, New South Wales
  - Sydney, New South Wales
  - Westmead, New South Wales
  - Nedlands, Western Australia
  - Parramatta
- Austria (2):
  - Vienna, Vienna
  - Vienna
- Canada (8):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - London, Ontario
  - Mississauga, Ontario
  - Montreal, Quebec
  - Sherbrooke, Quebec
- Chile (4):
  - Osorno, Los Lagos Region
  - Metropolitana, Santiago Metropolitan
  - Santiago, Santiago Metropolitan
  - Vitacura, Santiago Metropolitan
- Bogotá, Bogota D.C., Colombia
- Czechia (2):
  - Hradec Králové
  - Prague
- France (3):
  - Paris, Cedex 12
  - Boredaux
  - Lyon
- Germany (10):
  - Tübingen, Baden-Wurttemberg
  - München, Bavaria
  - Hamburg, Hamburg
  - Bonn, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Dresden, Saxony
  - Leipzig, Saxony
  - Berlin, State of Berlin
- Hong Kong (2):
  - Hong Kong
  - Kowloon
- Hungary (3):
  - Budapest
  - Debrecen
  - Pécs
- Israel (10):
  - Afula
  - Beersheba
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Tel Aviv
  - Ẕerifin
- Italy (9):
  - Udine, Friuli Venezia Giulia
  - Rome, Lazio
  - Milan, Lombardy
  - Florence, Tuscany
  - Padua, Veneto
  - Ancona
  - Bologna
  - Milan
  - Sassari
- Japan (16):
  - Inba-gun, Chiba
  - Fukuoka, Fukuoka
  - Miyako-gun, Fukuoka
  - Sapporo, Hokkaido
  - Himeji, Hyōgo
  - Yamato, Kanagawa
  - Yokohama, Kanagawa
  - Kumamoto, Kumamoto
  - Iga, Mie-ken
  - Nagasaki, Nagasaki
  - Nara, Nara
  - Osaka, Osaka
  - Chōfu, Tokyo
  - Itabashi-ku, Tokyo
  - Ōta-ku, Tokyo
  - Taito-ku, Tokyo
- Slovakia (4):
  - Bratislava
  - Ružomberok
  - Trenčín
  - Žilina
- South Korea (4):
  - Seongnam-si, Gyeonggido
  - Busan
  - Incheon
  - Seoul
- Spain (9):
  - Albacete, Albacete
  - Barcelona, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - San Cugat Del Vallès, Barcelona
  - Seville, Sevilla
  - Valencia, Valencia
  - Valladolid, Valladolid
  - Barakaldo, Vizcaya
  - Valencia
- Switzerland (3):
  - Bern, Canton of Bern
  - Zurich, Canton of Zurich
  - Lausanne

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 27 centers, between 10 October 2014 (first subject first visit) and 17 June 2015 (last subject last visit).
Pre-assignment Details: Study was planned to be conducted in 2 parts, Part A and B, in Part A 89 subjects were enrolled, of them 37 were screen failure and 52 were assigned to treatment, 1 subject was excluded from all analysis sets due to protocol deviations and 51 subjects were analyzed. Part B was not initiated and the study terminated following completion of Part A.
Groups:
- Part A Regorafenib: Participants self-administered 30 milligram per milliliter (mg/mL), 25 microliter (mcL),1 drop of Regorafenib eye drops, topically thrice daily (TID) to the study eye for 12 weeks.
Period: Overall Study
Arm/Group | Part A Regorafenib
Started | 52
Treated and Valid for Full Analysis Set | 51
Completed | 48
Not Completed | 4
Not completed — Death | 1
Not completed — Other reasons | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Part A Regorafenib
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) as Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) Letter Score at Study Week 4 for Study Part A
Description: Participants will be assessed at each clinic visit for best corrected visual acuity using the early treatment diabetic retinopathy study chart. Visual function of the study eye and the fellow eye was assessed using the ETDRS. The participant's ETDRS testing score was recorded in the appropriate eCRF page at each study visit. For participants that dropped out or received rescue treatment the last observation before drop-out or administration of rescue treatment was carried forward. A higher score represents better functioning.
Time Frame: Baseline, Week 4
Population: Full Analysis Set (FAS): included participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Part A Regorafenib
Number analyzed (Participants) | 50
Score on scale | 1.18 (7.55) [lower limit 7.55]

2. Primary Outcome: Change From Baseline in BCVA as Measured by ETDRS Letter Score at Study Week 12 for Study Part A
Description: Participants were assessed at each clinic visit for best corrected visual acuity using the early treatment diabetic retinopathy study chart. Visual function of the study eye and the fellow eye was assessed using the ETDRS protocol. ETDRS testing score was recorded in the appropriate eCRF page at each study visit. For participants that dropped out or received rescue treatment the last observation before drop-out or administration of rescue treatment was carried forward. A higher score represents better functioning.
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS): included subjects who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Part A Regorafenib
Number analyzed (Participants) | 50
Score on scale | -2.36 (7.68) [lower limit 7.68]

3. Secondary Outcome: Percentage of Participants With Individual Changes in BCVA of Greater Than Equal to (>=) 0 Letters of Vision From Study Week 4 to Week 12 for Study Part A
Description: Participants were assessed at each clinic visit for BCVA using the early treatment diabetic retinopathy study chart. For participants that dropped out or received rescue treatment the last observation before drop-out or administration of rescue treatment was carried forward.
Time Frame: Week 4, Week 12
Population: Full Analysis Set (FAS): included subjects who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Part A Regorafenib
Number analyzed (Participants) | 50
percentage of participants | 42

4. Secondary Outcome: Percentage of Participants With a Loss in BCVA of >= 10 Letters From Baseline to Study Week 12 for Study Part A
Description: as for outcome 3
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS): included subjects who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Part A Regorafenib
Number analyzed (Participants) | 50
percentage of participants | 16

ADVERSE EVENTS:
Time Frame: From the start of study treatment until 30 days after last dose of study drug treatment (up to Week 16).
Groups:
- Part A Regorafenib: Participants self-administered 30 mg/mL, 25 mcL, 1 drop of regorafenib eye drops, topically thrice daily (TID) to the study eye for 12 weeks.
Arm/Group | Part A Regorafenib
Serious Adverse Events (participants affected / at risk) | 3/51
Other Adverse Events (participants affected / at risk) | 11/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Regorafenib (N=51)
Acute myocardial infarction (Cardiac disorders) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Visual acuity tests abnormal (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Regorafenib (N=51)
Visual acuity reduced (Eye disorders) | 6
Visual acuity tests abnormal (Investigations) | 5

LIMITATIONS AND CAVEATS:
As the study was prematurely terminated since pre-defined proof of concept (PoC) criteria were not met in Part A, hence part B was not initiated. Part B related end points and data were not reported since it is not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In mulit centre studies result of study are to be published only through coordination by Bayer in order to combine the results of all centres. Center free to publish its results provided the overall results have not been published within 18 months from study completion (data base lock), subject to the compliance to remaining terms set forth in the PI contract.